CLINICAL TRIAL: NCT04378400
Title: An Institutional Audit of the Short Term Complications and Long Term Outcomes of Patients Undergoing Laparoscopic Sacrocolpopexy for Vault/cervical Prolapse.
Status: Enrolling by invitation | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Jan Deprest, MD, PhD, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S63523
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Vault Prolapse, Vaginal
Keywords: sacropexy; audit
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Sacrocolpopexy — Sacrocolpopexy is offered to patients with symptomatic prolapse (≥stage II) of the vaginal apex (vault or cervix). The procedure involves dissection of the promontory and the vaginal vault, suturing of two meshes to the anterior and posterior aspect of the vagina using minimally three rows of sutures on each side, and one row at the apex. Thereafter the mesh is fixed with staples to the promontory and the peritoneum closed, with staples and a running suture.

SUMMARY:
An institutional audit of the short term complications and long term outcomes of patients undergoing laparoscopic sacrocolpopexy for vault/cervical prolapse.

DETAILED DESCRIPTION:
The aim of this study is to audit the outcomes of laparoscopic sacrocolpopexy procedures done in our unit. The investigators aim to permanently monitor outcomes of this procedure correcting vaginal vault prolapse or cervical descent. Auditing institutional performance with pelvic floor procedures is increasingly being required by (inter)national societies in pelvic floor medicine, so that patients can be counseled on outcomes they can expect at a given institution.

Sacrocolpopexy is offered to patients with symptomatic prolapse (≥stage II) of the vaginal apex (vault or cervix). The procedure involves dissection of the promontory and the vaginal vault, suturing of two meshes to the anterior and posterior aspect of the vagina using minimally three rows of sutures on each side, and one row at the apex. Thereafter the mesh is fixed with staples to the promontory and the peritoneum closed, with staples and a running suture.

The investigators started auditing this procedure 20 years ago because of the conversion to laparoscopy.

High anatomical and subjective cure rates are reported on the medium term (range 12-60 months), though long-term data (60 months or longer) are scarce and most studies focus on anatomical outcomes.4 The investigators recently published medium term outcomes of patients operated up to 2014 1. Now the aim is to extend this audit to patients operated since 2014 and install a process of permanent monitoring our performance with this operation. The investigators also want to use the availability of outcomes in large numbers and/or the long term, to detect potential rare or long term complications, and study the effects of small technical increments such as extending dissections, associate other pelvic floor reconstructive procedures or the change in bio-materials used for this operation. All these may affect outcome.

Primary outcome is a subjective outcome, using a patient-centered approach and report patient reported out-comes. Additional outcomes such as anatomical failure, or complications, both by occurrence and time point, re-interventions, and pelvic floor functional outcomes are secondary outcomes that allows the investigators to benchmark their performance to previous studies and other series. Key in an objective assessment process is that patients are examined by an experienced clinician not involved in the management, which will also be used herein.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, female subjects must meet the following inclusion criteria:

1. Having undergone laparoscopic sacrocolpoexy at our unit.
2. Agreeing to participate in the study, including completion of study-related procedures, evaluations and questionnaires, and giving informed consent.
3. Follow up period of at least 6 months since the operation.

Exclusion Criteria:

None apart from not meeting the above criteria

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Since our last audit (April 30, 2014), we have operated on more than probably another 250 patients, who will be contacted. Based on our previous experience, we expect a 85% response rate.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Subjective Success Rate | Up to 10 years postoperative
  Subjective Success assessed by the Patient Global Impression of Change (PGI-C) tool, which is a 5-point Likert scale, where the patients are asked the following question at the follow up visit: "Compared with how you were doing before your recent pelvic floor operation, would you say that now you are: "much better", "a little better", "about the same", "a little worse" or "much worse".

SECONDARY OUTCOMES:
Objective success | Up to 10 years postoperative
  Objective Success will be defined as: achievement of a POP-Q score Stage ≤1, without re-intervention for POP or graft related complication at approximately 12 months.
Postoperative complications | Up to 10 years postoperative
  Occurrence of operative complications: classified as either intra-operative or postoperative (within 3 months of operation), and according to the Dindo classification, as we earlier did.
Reintervention rate | Up to 10 years postoperative
  Reintervention for prolapse as well as its compartment, at any time point during follow up. The time point of reintervention will be a variable per se.
Postoperative graft related complications (GRC) | Up to 10 years postoperative
  Postoperative graft related complications (GRC) out of a (non-limitative) list of de novo dyspareunia, worsening of pre-existing dyspareunia, incidence of chronic pain, occurrence of exposure, extrusion or any other complication and any reintervention because of the above. GRC will be categorized according to the IUGA classification
Prolapse Quality of Life (P-QoL) | Up to 10 years postoperative
  P-QoL: self-reported severity of symptoms in patients with urogenital prolapse and their impact on 9 different quality of life domains with scores for each domain, ranging between 0 and 100. Higher scores indicate a greater impairment of quality of life. This has been validated for the Flemish population

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Page AS, Cattani L, Pacquee S, Claerhout F, Callewaert G, Housmans S, Van der Aa F, D'Hoore A, Deprest J. Long-term Data on Graft-Related Complications After Sacrocolpopexy With Lightweight Compared With Heavier-Weight Mesh. Obstet Gynecol. 2023 Jan 1;141(1):189-198. doi: 10.1097/AOG.0000000000005021. Epub 2022 Nov 30. PMID 36701619